CLINICAL TRIAL: NCT03831048
Title: Clinical Trial to Evaluate the Safety and Effectiveness of The Portable Organ Care System (OCS™) Heart For Resuscitation, Preservation and Assessment of Hearts From Donors After Circulatory Death (DCD Heart Trial)
Brief Title: Donors After Circulatory Death Heart Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCS-CAR-03202019
Record Dates: First submitted 2019-01-22; First posted 2019-02-05 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2022-12

CONDITIONS: Heart Transplant
Keywords: Heart preservation; Beating heart transplant
MeSH Terms: interventions — Cryopreservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- DCD Heart Possible (Experimental)
  Interventions: Device: OCS Heart System
- Standard of Care Heart Only (Active Comparator)
  Interventions: Other: Cold Storage

INTERVENTIONS:
Device: OCS Heart System — Preserving and assessing donor after circulatory death hearts for transplant
  Arms: DCD Heart Possible
Other: Cold Storage — Active comparator intervention
  Arms: Standard of Care Heart Only

SUMMARY:
To evaluate the effectiveness of the OCS Heart System to resuscitate, preserve and assess hearts donated after circulatory death for transplantation to increase the pool of donor hearts available for transplantation.

DETAILED DESCRIPTION:
A prospective, randomized and concurrent controlled, non-inferiority pivotal trial in which subjects who receive a DCD donor heart transplant will be compared to subjects who receive a standard criteria donor heart transplant (Standard of Care 1 [SOC1] and Standard of Care 2 [SOC2] - from both randomized and concurrent control groups), adjusting for differences in risk factors.

ELIGIBILITY:
Donor Inclusion

* Maastricht Category III DCD donor, defined as expected death after the withdrawal of life- supportive therapy (WLST)
* Donor age 18-49 years old inclusive
* Warm ischemic time (WIT) ≤ 30 mins, with warm ischemic time defined as: Time from when mean systolic blood pressure (SBP) is < 50 mmHg or peripheral saturation < 70% to aortic cross-clamp and administration of cold cardioplegia in the donor.

Donor Exclusion

* Previous cardiac surgery
* Known coronary artery disease
* Cardiogenic shock or myocardial infarction, or
* Sustained terminal ejection fraction (EF) of ≤ 50%, or
* Significant valve disease except for competent bicuspid aortic valve

Recipient Inclusion

* Primary heart transplant candidates
* Age ≥ 18 years old
* Signed: (1) written informed consent document; (2) authorization to use and disclose protected health information; and (3) consent to TransMedics' use of recipients' United Network for Organ Sharing (UNOS)/Organ Procurement and Transplantation Network (OPTN) data and recipients' Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) data.

Recipient Exclusion

* Prior solid organ or bone marrow transplant
* Chronic use of hemodialysis or diagnosis of chronic renal insufficiency
* Multi-organ transplant
* Investigator unwilling to randomize to either arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - University of California San Diago, La Jolla, California
  - Cedars Sinai, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - AdventHealth, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - St. Vincent Cardiovascular Research Institute, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nyph/Cumc, New York, New York
  - Montefiore, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Duke University, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Sentara, Norfolk, Virginia
  - Virgina Commonwealth University, Richmond, Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Merani S, Urban M, Westphal SG, Dong J, Miles CD, Maskin A, Hoffman A, Langnas AN. Improved Early Post-Transplant Outcomes and Organ Use in Kidney Transplant Using Normothermic Regional Perfusion for Donation after Circulatory Death: National Experience in the US. J Am Coll Surg. 2024 Jan 1;238(1):107-118. doi: 10.1097/XCS.0000000000000880. Epub 2023 Sep 29. PMID 37772721
- [Derived] Schroder JN, Patel CB, DeVore AD, Bryner BS, Casalinova S, Shah A, Smith JW, Fiedler AG, Daneshmand M, Silvestry S, Geirsson A, Pretorius V, Joyce DL, Um JY, Esmailian F, Takeda K, Mudy K, Shudo Y, Salerno CT, Pham SM, Goldstein DJ, Philpott J, Dunning J, Lozonschi L, Couper GS, Mallidi HR, Givertz MM, Pham DT, Shaffer AW, Kai M, Quader MA, Absi T, Attia TS, Shukrallah B, Sun BC, Farr M, Mehra MR, Madsen JC, Milano CA, D'Alessandro DA. Transplantation Outcomes with Donor Hearts after Circulatory Death. N Engl J Med. 2023 Jun 8;388(23):2121-2131. doi: 10.1056/NEJMoa2212438. PMID 37285526
- [Derived] Shudo Y, Benjamin-Addy R, Koyano TK, Hiesinger W, MacArthur JW, Woo YJ. Donors after circulatory death heart trial. Future Cardiol. 2021 Jan;17(1):11-17. doi: 10.2217/fca-2020-0070. Epub 2020 Jul 6. PMID 32628044

RESULTS

PARTICIPANT FLOW:
Groups:
- DCD Heart: OCS Heart System: Preserving and assessing donor after circulatory death hearts for transplant
- Standard of Care Heart: Cold Storage: Active comparator intervention
Period: Overall Study
Arm/Group | DCD Heart | Standard of Care Heart
Started | 90 | 90
Per Protocol Population | 80 | 86
Completed | 76 | 75
Not Completed | 14 | 15
Not completed — Protocol Violation | 9 | 3
Not completed — Death | 4 | 9
Not completed — Re-transplant | 0 | 2
Not completed — Protocol violation and death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DCD Heart | Standard of Care Heart | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] — Recipient age
  years | 51.3 (12.6) | 55 (11.4) | 52.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Recipient sex
  Participants
    Female | 24 | 24 | 48
    Male | 66 | 66 | 132
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 20 | 48
  White | 62 | 66 | 128
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Patient survival 6 months post-transplant
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | DCD Heart | Standard of Care Heart
Number analyzed (Participants) | 80 | 86
Participants | 76 | 75
Statistical Analysis 1: Comparison: DCD Heart vs Standard of Care Heart; The null and alternative hypotheses for the primary endpoint are as follows: H0: pSOC - pDCD ≥ 0.20 vs. H1: pSOC - pDCD < 0.20 where pDCD and pSOC represent the true survival proportions at the six months follow-up visit for DCD and SOC heart transplant patients, respectively; Test type: Non-Inferiority — The primary analysis of this endpoint will be performed using a linear probability model, with the following terms in the model: (1) treatment; and (2) the known donor and recipient risk factors listed above. Variables that make the model fail to converge will be dropped from the model. The test will be conducted at the one-sided 0.05 level of significance; p < 0.0001, Regression, Linear — No multiple comparison adjustment; Mean Difference (Final Values) = -0.032, 90% CI 2-sided [-0.098 to 0.034]

2. Secondary Outcome: Utilization Rate
Description: Utilization Rate, defined as the number of eligible DCD donor hearts that met the warm ischemic time limit above and were instrumented on the OCS Heart System that meet the acceptance criteria for transplantation after OCS Heart preservation divided by the total number of eligible DCD donor hearts that met the warm ischemic time limit above and were instrumented on the OCS Heart System.
Time Frame: Within 24 hours post-transplant
Population: Per protocol, Analysis Population includes DCD donor hearts that met the warm ischemic time limit, then were instrumented on OCS Heart System and transplanted.
  The utilization rate is analyzing only the number of hearts instrumented/transplanted, and not number of participants.
Measure: Count of Units; unit: Hearts Instrumented
Units Other Than Participants: Hearts Instrumented
Groups:
- OCS Heart Instrumentation: Total hearts instrumented on OCS
Arm/Group | OCS Heart Instrumentation
Number analyzed (Participants) | 80
Number analyzed (Hearts Instrumented) | 91
Hearts Instrumented | 80
Statistical Analysis 1: Comparison: OCS Heart Instrumentation; No null hypothesis test; Test type: Other — No hypothesis test; No statistical hypothesis testing. This endpoint will be summarized for the OCS Heart Population using counts and percentages and an exact (Clopper-Pearson) 95% confidence interval for the true percentage based on the binomial distribution. It will also be summarized for the modified OCS Heart Population, defined as the number of DCD hearts that were successfully transplanted after preservation and assessment on the OCS divided by the total number of DCD donor hearts that were instrumented on the OCS

ADVERSE EVENTS:
Time Frame: Per the protocol, all SAEs will be collected for the first 30 days post-transplant for the DCD Heart Transplanted Recipients group only. All-Cause Mortality was assessed for 6 months post-transplant as reported.
Description: Per the protocol, only serious adverse events (SAEs) and Heart Graft-Related SAE's (HGRSAEs) will be captured in this study for the DCD Heart Transplanted Recipients group.
  SAEs and HGRSAEs will not be captured for the Standard of Care Heart Transplanted Recipient group.
Arm/Group | DCD Heart | Standard of Care Heart
All-Cause Mortality (participants affected / at risk) | 5/90 | 10/90
Serious Adverse Events (participants affected / at risk) | 67/90 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCD Heart (N=90) | Standard of Care Heart (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | NA
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | NA
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | NA
Atrial fibrillation (Cardiac disorders) | 1 (1) | NA
Atrial flutter (Cardiac disorders) | 1 (1) | NA
Cardiac arrest (Cardiac disorders) | 1 (1) | NA
Cardiac tamponade (Cardiac disorders) | 2 (2) | NA
Cardiogenic shock (Cardiac disorders) | 2 (2) | NA
Left ventricular dysfunction (Cardiac disorders) | 16 (16) | NA
Pericardial effusion (Cardiac disorders) | 4 (4) | NA
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | NA
Right ventricular dysfunction (Cardiac disorders) | 6 (6) | NA
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | NA
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | NA
Diarrhoea (Gastrointestinal disorders) | 1 (1) | NA
Gastrointestinal necrosis (Gastrointestinal disorders) | 2 (2) | NA
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | NA
Volvulus (Gastrointestinal disorders) | 1 (1) | NA
Transplant rejection (Immune system disorders) | 18 (18) | NA
Bacteraemia (Infections and infestations) | 2 (2) | NA
Endocarditis (Infections and infestations) | 1 (1) | NA
Fungal infection (Infections and infestations) | 1 (1) | NA
Nasopharyngitis (Infections and infestations) | 1 (1) | NA
Pneumonia (Infections and infestations) | 5 (5) | NA
Sepsis (Infections and infestations) | 2 (2) | NA
Iatrogenic injury (Injury, poisoning and procedural complications) | 1 (1) | NA
Traumatic haemothorax (Injury, poisoning and procedural complications) | 2 (2) | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Brain hypoxia (Nervous system disorders) | 1 (1) | NA
Ischaemic stroke (Nervous system disorders) | 1 (1) | NA
Migraine (Nervous system disorders) | 1 (1) | NA
Seizure (Nervous system disorders) | 2 (2) | NA
Spinal stroke (Nervous system disorders) | 1 (1) | NA
Delirium (Psychiatric disorders) | 2 (2) | NA
Acute kidney injury (Renal and urinary disorders) | 15 (15) | NA
Renal failure (Renal and urinary disorders) | 4 (4) | NA
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | NA
Deep vein thrombosis (Vascular disorders) | 2 (2) | NA
Deep vein thrombosis (Vascular disorders) | 1 (1) | NA
Haemorrhage (Vascular disorders) | 10 (10) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT03831048/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT03831048/SAP_001.pdf